CLINICAL TRIAL: NCT01552798
Title: A Double-Blind, Randomized, Parallel, Placebo-Controlled Trial Assessing the Analgesic Efficacy of a Single Dose of Fast Release Aspirin 1000 mg and Acetaminophen 1000 mg in Tension Type Headache Pain
Brief Title: Efficacy of a Single Dose of Aspirin vs. Acetaminophen in Tension Type Headache
Acronym: Tarot Headache
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15771
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Aspirin; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAY1019036)
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetaminophen
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAY1019036) — 2 x 500 mg fast release aspirin tablets (1000 mg) and 2 x placebo acetaminophen caplets
  Arms: Arm 1
Drug: Acetaminophen — 2 x 500 mg acetaminophen caplets (1000 mg) and 2 x placebo fast release aspirin tablets
  Arms: Arm 2
Drug: Placebo — 2 x placebo acetaminophen caplets and 2 x placebo fast release aspirin tablets
  Arms: Arm 3

SUMMARY:
The purpose of this trial is to determine if a single, oral dose of a fast release aspirin 1000 mg provides relief compared to acetaminophen 1000 mg and placebo in subjects with tension-type headache pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers ages 18-65 years old
* History of an onset of tension type headaches before age 50
* Experiencing over the last year ≥ 4 tension type headaches of at least moderate intensity per month and with the majority of headaches lasting greater than three hours, that meet commonly recognized criteria for diagnosis per the International Headache Society
* History of response to treatment with over-the-counter (OTC) analgesics
* Understand the pain rating scales (as judged by the trial coordinator)
* Present with at least moderate headache pain on a 0-10 point numerical rating scale (a score of at least 4 on an 11 point scale ranging from 0 to 10) at the Treatment Visit
* Onset of pain within three hours of the Treatment Visit
* Confirmation by a physician of acute tension type headache symptoms as described by the International Headache Society diagnostic criteria

Exclusion Criteria:

* History of hypersensitivity to aspirin, salicylates, other NSAIDs, acetaminophen, and similar pharmacological agents or components of the investigational products, including the placebo
* Use of any immediate release analgesic/anti-pyretic within four hours or use of any sustained release or long acting analgesic/anti-pyretic within 12 hours proceeding administration of Investigational Product
* Presence of symptoms that are consistent with menstrual headache or migraine headache as described by the International Headache Society diagnostic criteria
* History of migraine headaches more than once per month
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than 50 percent obstruction (polyposis nasi, marked septal deviation) that can interfere with the conduct of the trial in the judgment of the Investigator
* Current or past history of bleeding disorder(s)
* History of gastrointestinal bleeding or perforation, related to previous Nonsteroidal Anti-inflammatory Drugs (NSAID) therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Recent head or neck trauma (within 2 weeks)
* Current use of blood thinning (anticoagulant), low dose aspirin, or steroid drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03-12 (Actual); Primary Completion 2012-06-04 (Actual); Study Completion 2012-06-04 (Actual)

PRIMARY OUTCOMES:
Time to meaningful pain relief (defined as the time when the subject indicates pain relief that is meaningful to the subject) | Up to 2 hours post-dose

SECONDARY OUTCOMES:
Time to first perceptible relief | Up to 2 hours post-dose
  Is defined as the time when the subject presses the first stopwatch
Time to first perceptible relief confirmed | Up to 2 hours post-dose
  The subjects would meet this outcome if they answer "yes" when asked directly after stopping the first stopwatch, if they marked a "1" on the relief pain scale or if they stopped the 2nd stop watch.
Change from baseline in pain intensity score at different time points (on an 11-point Categorical Pain Intensity Scale, 0 = no pain, 10 = severe pain) | At baseline, 30, 60, 90 and 120 minutes post-dose, and immediately prior to the use of any rescue medication
Pain Relief on 5-point Categorical Scale (0 = no relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, and 4 = complete relief) | At 30, 60, 90 and 120 minutes post-dose, and immediately prior to the use of any rescue medication
Summed time weighted of Pain Intensity Differences (PID) scores over first hour (SPID0-1) | Up to 1 hour
Summed time weighted of Pain Intensity Differences (PID) scores over 2 hours (SPID0-2) | Up to 2 hours
Summed time weighted total pain relief scores over first hour (TOTPAR0-1) | Up to 1 hour
Summed time weighted of Total Pain Relief Scores (TOTPAR) scores over 2 hours (TOTPAR0-2) | Up to 2 hours
Summed, time weighted of Pain Relief and Pain Intensity Differences (PID) over first hour (SPRID0-1) | Up to 1 hour
Summed, time weighted of Pain Relief and Pain Intensity Differences (PID) over 2 hours (SPRID0-2) | Up to 2 hours
Time to first intake of rescue medication | Up to 2 hours
Cumulative proportion of subjects taking rescue medication by time point | Up to 2 hours
Global assessment of the investigational product as a pain reliever: 0 = poor, 1 = fair, 2 = good, 3 = very good or 4 = excellent | At 2 hours post-dose or immediately before the first intake of rescue medication, whichever is earlier
Safety variable will be summarized using descriptive statistic based on adverse events collection | Up to 5 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Westside Family Medical Center, Kalamazoo, Michigan, United States